CLINICAL TRIAL: NCT02236936
Title: Randomized Phase III Study: Supplemental Parenteral Nutrition for Patients With Locally Advanced Inoperable Tumors of the Head and Neck, Receiving Definitive Radiotherapy With Cetuximab or Cisplatin
Brief Title: Parenteral Nutrition for Patients Treated for Locally Advanced Inoperable Tumors of the Head and Neck
Acronym: AGMT_HNO_PN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to low recruitment
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_HNO_PN
Record Dates: First submitted 2014-09-05; First posted 2014-09-11 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Squamous Cell Carcinoma of the Hypopharynx Stage III; Squamous Cell Carcinoma of the Hypopharynx Stage IV; Laryngeal Squamous Cell Carcinoma Stage III; Laryngeal Squamous Cell Carcinoma Stage IV; Oropharyngeal Squamous Cell Carcinoma Stage III; Oropharyngeal Squamous Cell Carcinoma Stage IV; Squamous Cell Carcinoma of the Oral Cavity Stage III; Squamous Cell Carcinoma of the Oral Cavity Stage IV; Locally Advanced Malignant Neoplasm
Keywords: Squamous Cell Carcinoma; Head and neck; SCCHN; Parenteral nutrition; Larynx; Hypopharynx; Cavum oris; Radiotherapy; Cetuximab; Cisplatin
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Hyperphagia; Laryngeal Diseases | interventions — Emulsions; Cetuximab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Standard of care (Active Comparator): Standard care of parenteral nutrition (with or without parenteral nutrition during radio-chemotherapy or radio-immunotherapy in combination with Cetuximab or Cisplatin.
  Concomitant radiotherapy and immunotherapy (radio-immunotherapy) with Cetuximab or concomitant radiotherapy and chemotherapy (radio-chemotherapy) with Cisplatin
  Interventions: Dietary Supplement: Standard care of parenteral nutrition; Biological: Cetuximab; Drug: Cisplatin; Radiation: Radiotherapy
- Arm B - Parenteral over night nutrition (Experimental): Parenteral over night nutrition with ZentroOLIMEL 5.7% parenteral over night with electrolytes, vitamins (Cernevit®) and micronutrients (Addel Trace® or Nutryelt®) 15 ml/kg body weight/day (weight loss >5% from baseline; parenteral nutrition increased up to 25 ml/kg body weight per day) during radio-chemotherapy or radio-immunotherapy in combination with Cetuximab or Cisplatin.
  Concomitant radiotherapy and immunotherapy (radio-immunotherapy) with Cetuximab or concomitant radiotherapy and chemotherapy (radio-chemotherapy) with Cisplatin
  Interventions: Dietary Supplement: Parenteral over night nutrition; Biological: Cetuximab; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Dietary Supplement: Standard care of parenteral nutrition — Standard treatment according to the discretion of the center, any required nutritional support (enteral tube feeding by nasogastric tube or percutaneous endoscopic gastrostomy) when considered necessary is allowed
  Other Names: PN
  Arms: Arm A - Standard of care
Dietary Supplement: Parenteral over night nutrition — Patients in interventional Arm B will receive parenteral overnight nutrition with ZentroOLIMEL® 5.7% with electrolytes, vitamins (Cernevit®) and micronutrients (Addel Trace® or Nutryelt®) starting with 15 ml/kg body weight/day. In case of weight loss of more than 5%, dose of ZentroOLIMEL® has to be increased up to 25 ml/kg/body weight/day.
  Other Names: Emulsion for infusion
  Arms: Arm B - Parenteral over night nutrition
Biological: Cetuximab — Weekly during radiotherapy; not given if cisplatin is given during radiotherapy
  Cetuximab 400 mg/m2 (saturation) Cetuximab 250mg/m2 (during radiotherapy; in total 7x)
  Other Names: Erbitux
Drug: Cisplatin — Cisplatin total dose of >200 mg administered weekly (40 mg/m2/week) or every three weeks (100 mg/m2 every three weeks) according to local standard; not given in combination with cetuximab
  Other Names: Cisplatinum; CDDP
Radiation: Radiotherapy — 70 Gy / 5 fractions per week, over 7 weeks
  Other Names: RTX

SUMMARY:
Prevention of critical weight loss. In patients with Squamous Cell Carcinoma of the Head and Neck (SCCHN) weight loss is a relevant clinical problem during radiotherapy and might result in higher treatment related toxicity and discontinuation of a potential curative treatment. Thus the investigators want to evaluate the efficacy of overnight parenteral nutritional (PN) support in patients with SCCHN treated with curative radiotherapy (RTX) in combination with Cetuximab (E) or Cisplatin (P).

DETAILED DESCRIPTION:
The investigators hypothesize that about 60% of patients receiving RTX without supplemental PN will suffer from critical weight loss of more than 5% during treatment - supplemental overnight PN might result in significant improvement of the nutritional status .

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is eligible for definitive curative radio-chemotherapy with Cisplatin or radio-immunotherapy with Cetuximab.
* Written informed consent obtained prior to any study specific screening activities and patients have to be able to comply with this protocol.
* Histologically confirmed local advanced squamous cell carcinoma of the Larynx, Hypopharynx, Oropharynx or Cavum oris treated with definitive radiotherapy in combination with Cisplatin or Cetuximab.
* p16 status available
* Age ≥ 18
* Women of childbearing potential must have a negative pregnancy test at screening and must use effective contraception.

Exclusion Criteria:

* Distant metastases
* Prior radiation (Head and neck area)
* Pregnant or lactating women
* History of other malignancy; yet patients who have been disease-free for 5 years or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent other cancer therapy (chemotherapy, immunotherapy, antihormonal or biologic therapy) or concurrent treatment with an investigational drug.
* Serious medical or psychiatric disorders that would interfere with the patient's safety or informed consent.
* Participation in another interventional clinical study at time of study inclusion (except follow-up period without treatment for more than 30 days) or denial of the simultaneous participation in a non-interventional study by the PI of the study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Loss of body weight by more than 5% at the end of radiotherapy | Difference between baseline and week 8 (after end of RTX)
  Weekly body weight assessments - standardized method for all study sites

SECONDARY OUTCOMES:
Bioelectrical Impedance Analysis (BIA): reduction of phase angle by > 10% during treatment/observation | Prior to and 1 year after start of RTX, within 7 days and 3 months after end of RTX
  Determination of parameters on functional nutritional status: fat-free mass (FFM), total body water (TBW), body fat and phase angle will be evaluated by BIA

OTHER OUTCOMES:
Assessment of physical strength | Prior to RTX, weekly during RTX, within 1 week and 3 months after end of RTX
  Handgrip strength measurement, mean value of three consecutive measurements
Number of implanted PEG tubes | From start of RTX until 3 months after end of RTX
  The number of implanted PEG tubes will be recorded
Acute toxicity during radiotherapy | During 7 weeks of radiotherapy, at end of radiotherapy and 3 months after radiotherapy
  Acute toxicity according to Common Terminology Criteria for Adverse Events (CTCAE 4.0.)
Chronic toxicity after treatment | 3 months after end of radiotherapy
  Chronic toxicity evaluated according to RTOG (Radiation Therapy Oncology Group)/EORTC (European Organisation for Research and Treatment of Cancer) - Toxicity Criteria
Dose and dose intensity of radiotherapy | At start and end of radiotherapy (duration of radiotherapy 7 weeks)
  Dose and dose intensity including delay of scheduled therapy and absolute dose of radiotherapy applied.
Progression-free (PFS) | From start until 3 months after end of RTX
  The study will be finished one year post RTX and clinical al data on PFS will be obtained. In addition, patient will be asked to agree to collection of information regarding PFS even after completion of the trial.
Overall survival (OS) | From start until 3 months after end of RTX
  The study will be finished one year post RTX and clinical data on OS will be obtained. In addition, patient will be asked to agree to collection of information regarding OS even after completion of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Keil, Prof.Dr., Principal Investigator — Hanuschkrankenhaus
Locations (7):
- Austria (7):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universität Graz, HNO Universitätsklinik, Graz
  - Klinikum Klagenfurt am Wörthersee, HNO-Abteilung, Klagenfurt
  - Ordensklinikum Linz - Barmherzigen Schwestern, Abteilung f. HNO, Kopf- und Halschirurgie, Linz
  - Krankenhaus Hietzing, Sonderabteilung f. Strahlentheapie, Vienna
  - Hanuschkrankenhaus, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt

REFERENCES:
- See also: Sponsor — http://www.agmt.at